CLINICAL TRIAL: NCT01883037
Title: To Compare the Clinical Accuracy of Glucose Measurement During Oral Glucose Tolerance Test Using Two Methods: i) Laboratory Standard Technique, ii) HemoCue Glucose 201 RT System
Brief Title: Comparing Laboratory Blood Glucose Results With HemoCue Glucose 201 RT
Acronym: CFRD
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2012CF007B
Record Dates: First submitted 2013-06-13; First posted 2013-06-21 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Cystic Fibrosis related diabetes; Oral glucose tolerance test
MeSH Terms: conditions — Cystic Fibrosis | interventions — Blood Glucose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Laboratory blood glucose: Blood glucose value from Lab
  Interventions: Other: Blood glucose results
- HemoCue Glucose 201 RT: Blood glucose value from HemoCue Glucose 201 RT
  Interventions: Other: Blood glucose results

INTERVENTIONS:
Other: Blood glucose results — The glucose value from the HemoCue Glucose 201 RT will be compared with the Trust Laboratory value.
  Other Names: HemoCue Glucose 201 RT

SUMMARY:
There are very few studies comparing the accuracy, sensitivity and specificity of HemoCue glucose 201 RT system with the laboratory gold standard.

The incidence of cystic fibrosis related diabetes (CFRD) has risen significantly as patients' survival improves. Around 30% of all cystic fibrosis (CF) adult patients have CFRD. Early diagnosis of CFRD is important to slow the deterioration of lung function and nutritional status, both of which increase mortality.

The oral glucose tolerance test (OGTT) is the accepted method for detecting CFRD and the Cystic Fibrosis Trust guidelines recommend that patients with CF over the age of twelve years should be screened annually.

The World Health Organisation has pointed out that due to the absence of a more specific biological marker to define diabetes, plasma glucose estimation remains the basis of diagnostic criteria. WHO recommends that venous plasma glucose should be the standard method for measuring and reporting glucose concentration in blood. However, it has also recognised that there is a widespread use of capillary sampling. Although fasting values for venous and capillary plasma glucose are the same, in the nonfasting state capillary samples will give higher results than venous samples, and glucose values require conversion which can be problematic.

HemoCue Glucose 201 RT (HGS 201 RT) analyzer with plasma conversion provides laboratory quality test results at the point of care for the diagnosis, screening and monitoring of diabetes mellitus. The analyzer is easy to use and the system can be operated by nonlaboratory personnel, also the results can be presented immediately, leading to significant time and resource saving. The patient also benefits from having the result immediately instead of waiting for several hours. With immediate result, the doctor and health care professionals can provide education, support and reassurance, and implement care plans, if appropriate, at the earliest opportunity.

The aim of the study is to compare the clinical accuracy of HemoCue Glucose 201 RT with the laboratory standard method in the analysis of blood glucose concentration during oral glucose tolerance test.

DETAILED DESCRIPTION:
All CF patients attending annual review who require an OGTT will have a venous and a capillary blood sample taken simultaneously before (fasting = 0 min) and 2 hours (post glucose load = 120 min) after the administration of 75 grams Glucose solution orally.

The capillary sample will be analysed immediately using HGS 201 RT. The venous sample will be collected in a Fluoride Oxalate tube (WHO guideline) and sent to the Trust's laboratory for analysis as per usual practice.

ELIGIBILITY:
Inclusion Criteria:

The first 70 consecutive suitable consenting adult CF patients, who are 16 years of age and over, attending annual review at the Royal Brompton Hospital from June 2013 to March 2014, are eligible for the study

Exclusion Criteria:

Patients with an existing diagnosis of CFRD are exclude.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The first 70 consecutive adult CF patients, without cystic fibrosis related diabetes, who are 16 years of age and over, attending annual review at the Royal Brompton Hospital from June 2013, are eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Does HemoCue Glucose 201 RT provide lab-quality results in the analysis of glucose values during oral glucose tolerance tests? | One year
  The glucose value from the HemoCue Glucose 201 RT will be compared with the Trust Laboratory value. The sensitivity, specificity and clinical significance will be calculated.

SECONDARY OUTCOMES:
Is HemoCue Glucose 201 RT method cost saving relative to the traditional laboratory method for analysing glucose values taken during oral glucose tolerance tests? | One year
  The cost of using the HemoCue Glucose 201 RT will be compared with Trust Laboratory cost for analysing the glucose value from OGTT.

OTHER OUTCOMES:
2. To see if the HemoCue Glucose 201 RT offers sufficient advantages to make it a viable alternative to conventional testing | One year
  If using HemoCue Glucose 201 RT is shown to offer cost and clinical advantages over conventional testing then look to implement as standard test method and report more widely.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Simmonds, MD MRCP, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, United Kingdom